CLINICAL TRIAL: NCT03684369
Title: Improving Mobility and Reducing Fatigue in People With Multiple Sclerosis by Electrical Stimulation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project was not funded.
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other); Colorado State University (Other)
Responsible Party: Principal Investigator, Roger Enoka, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UColoradoBoulder2
Record Dates: First submitted 2018-08-24; First posted 2018-09-25 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: walking; balance; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented TENS (Experimental): Transcutaneous electrical nerve stimulation applied to each leg separately while participants perform steady submaximal contractions.
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Sham (Sham Comparator): Transient (10 s) application of transcutaneous electrical nerve stimulation applied to each leg separately while participants perform steady submaximal contractions .
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — Commercially available device will be used to apply weak electrical currents to arm and leg muscles in each of 18 treatment sessions.
  Other Names: Sham transcutaneous electrical nerve stimulation

SUMMARY:
The objective of the clinical trial is to quantify the capacity of a translatable protocol of electrical nerve stimulation (TENS) to improve walking performance and self-reported disabilities of persons with MS. The hypothesis is that activation of sensory nerve fibers with augmented TENS promotes recovery of sensorimotor function and improves the disability status of individuals with MS. The rationale for the proposed clinical trial is that the approach provides a low-cost therapeutic strategy for persons with MS to manage walking limitations and fatigue.

DETAILED DESCRIPTION:
The study will involve a randomized, double-blind, controlled trial. Randomization will be accomplished by recruiting two individuals with a similar level of disability at a time and flipping a coin (two persons present) to determine the group assignment (A or B) of the person who contacted the investigators first. The participants and outcome assessors will be blinded to group assignment. Both groups will receive the treatment (real or sham) during the first 4 weeks (3 sessions/week)and then there will be an 8-week follow-up period. Participants will be evaluated at weeks 0, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and speak English to ensure safe participation in the project
* Clinical diagnosis of multiple sclerosis
* Mild-to-moderate level of disability
* On stable doses of symptom-treating medications
* No MS exacerbations within the last 30 day
* Healthy enough to complete the protocol as indicated by the absence of a medical diagnosis or condition that is considered to be an absolute or relative contraindication to participating in tests that involve electrical nerve stimulation (e.g., not implanted devices or internal metal)
* Able to arrange own transportation to Boulder campus

Exclusion Criteria:

* Documented MS-related relapse within the last 30 days
* Medical diagnosis or condition that is considered to be a contraindication to participating in the intervention, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than basal cell cancer), other neurological disorders, or pregnancy.
* Vestibular disorder
* Musculoskeletal disorder
* History of seizure disorders
* >2 alcoholic drinks/day,or present history (last 6 months) of drug abuse
* Spasticity that requires the individual to change an activity more than once a week
* Skin disease or sensation problems in the legs or hands that influence some activities more than once a week
* Claustrophobia
* Metallic implants
* Inability to attend treatment sessions 3 days per week for 6 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Speed | Change from baseline at weeks 4, 8, and 12.
  Time to walk 25 ft as quickly as possible
Change in Walking Endurance | Change from baseline at weeks 4, 8, and 12
  Distance walked in 6 min when walking at a brisk pace
Change in Dynamic Balance | Change from baseline at weeks 4, 8, and 12
  Score achieved on the four components of the 14-item Mini-Balance Evaluation Systems Test (Mini-BESTest). The maximum score for each subscale are: anticipatory = 6, reactive postural control = 6, sensory orientation = 6, dynamic gait = 10. The subscales are added to provide a total score with a maximum of 28.
Change in Patient Determined Disease Steps | Change from baseline at weeks 4, 8, and 12
  A questionnaire with a self-assessment scale of disease status. The scores range from 0 = normal to 8 = bedridden.
Change in Modified Fatigue Impact Scale | Change from baseline at weeks 4, 8, and 12.
  A questionnaire that assesses the impact of fatigue experienced by persons with MS. Each of the 21 items is rated from 0 = Never to 5 = Almost always. The maximum total score = 105
Change in MS Walking Scale-12 | Change from baseline at weeks 4, 8, and 12.
  A 12-item, patient-rated measure of how much MS compromises walking ability. Each item is rated from 1 = Not at all to 5 = extremely. The maximum total score = 60.

SECONDARY OUTCOMES:
Change in Romberg Quotient | Change from baseline at weeks 4, 8, and 12.
  Ratio of the total sway area when standing with the eyes closed relative to that when the eyes are open. The test will be performed while standing on a firm surface and a foam surface.
Change Conditioned H-reflex Amplitude | Change from baseline at weeks 4, 8, and 12.
  Comparison of the percent reduction in the amplitude of the conditioned H-reflex amplitude in soleus while seated, standing with eyes open, and standing with eyes closed.
Change in Proprioception Tract | Change from baseline at weeks 4, 8, and 12.
  Change in MRI signal intensity in corticospinal tract
Change in Muscle Synergy Number | Change from baseline at weeks 4, 8, and 12
  Non-negative matrix factorization will be used to identify the number of muscle synergies when subjects walk on a treadmill.
Change in Force Steadiness | Change from baseline at weeks 4, 8, and 12.
  The coefficient of variation for force when subjects perform steady, submaximal contractions.
Change in Muscle Synergy TIming | Change from baseline at weeks 4, 8, and 12.
  The timing of the muscle synergies when subjects walk on a treadmill.
Change in Discharge characteristics | Change from baseline at weeks 4, 8, and 12.
  The mean and coefficient of variation for the times between action potentials during steady isometric contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Enoka, PhD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data obtained by individual participants.